CLINICAL TRIAL: NCT04122807
Title: Cryoablation of the Retrograde Fast Pathway as Treatment for AVNRT
Acronym: Cryo-FP
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114445
Record Dates: First submitted 2019-10-02; First posted 2019-10-10 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Atrioventricular Node Arrhythmia
Keywords: AVNRT; Cryoablation; PR interval
MeSH Terms: interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Prospective model with two groups based on PR interval on ECG, normal and prolonged PR
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mapping (Active Comparator): Standard treatment involving ablation of the slow pathway with cryotherapy
  Interventions: Procedure: Cardiac catheter ablation
- Ablation (Experimental): Mapping and ablation of the retrograde fast pathway with cryotherapy
  Interventions: Procedure: Cardiac catheter ablation

INTERVENTIONS:
Procedure: Cardiac catheter ablation — Cryoablation

SUMMARY:
In this study a new technique for ablation in atrioventricular nodal reentrant tachycardia using cryo-energy will be studied in cases where the standard approach has higher risk.

DETAILED DESCRIPTION:
Atrioventricular nodal reentrant tachycardia (AVNRT) is the most common cause of fast heartbeats in young people. People with AVNRT have two pathways within the heart, the fast pathway (FP) and slow pathway (SP). A treatment for AVNRT is ablation (burning or freezing) of the SP. This can be done with either radiofrequency or cryo-energy. A complication which occurs in 1% of cases is AV block (AVB), meaning the person needs a pacemaker.

Slow pathway ablation is a problem in people when the electrocardiogram (ECG) shows a long PR interval, with greater rates of AVB. This accounts for 5% of AVNRT cases. A possible solution is to treat the FP with cryo-energy and leave the SP intact. This pilot study aims to show this is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Documented supraventricular tachycardia (SVT)
* Planned to undergo electrophysiology (EP) study and ablation
* PR interval on ECG <220ms (Group 1) or >220ms (Group 2)

Exclusion Criteria:

* Pregnancy
* Age <18 years
* Inability to provide consent
* High likelihood of tachycardia mechanism other than AVNRT (e.g. Pre-excitation on surface ECG, atrial tachycardia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Termination of AVNRT | One day
  Number of participants where cryotherapy terminates AVNRT

SECONDARY OUTCOMES:
Freedom from recurrence | 1 year
  Number of participants with no recurrence of AVNRT during follow-up
Incidence of AV block | 1 year
  Number of participants where AV block is observed
Cardiac tamponade | 1 year
  Number of participants with pericardial effusion and/or tamponade following procedure
Vascular complications | 1 year
  Number of participants with groin hematoma or fistula requiring intervention following procedure

OTHER OUTCOMES:
Procedural time | Immediate
Fluoroscopy time | Immediate

CONTACTS AND LOCATIONS:
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No